CLINICAL TRIAL: NCT05860101
Title: An Investigation Into the Safety, Acceptability and Feasibility of a Brief Compassion-Focused Intervention for People Who Experience Distressing Mood Swings: A Case Series.
Brief Title: Compassion-Focused Therapy for Distressing Mood Swings: A Case Series
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Psychiatry, London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Tom Marsay, Trainee Clinical Psychologist, Institute of Psychiatry, London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R&D2022/059
Record Dates: First submitted 2023-04-25; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Bipolar Affective Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 week waitlist (Other)
  Interventions: Other: Compassion-Focused Therapy
- 2 week waitlist (Other)
  Interventions: Other: Compassion-Focused Therapy

INTERVENTIONS:
Other: Compassion-Focused Therapy — Compassion Focused Therapy (CFT) is based on the premise that we have three emotion regulation systems, the threat, drive and soothing systems. It has been suggested that our psychological wellbeing is dependent on maintaining a balance between these three systems, and if we lose this balance, e.g. the threat or drive systems become more dominant, then we start to experience emotional difficulties (Gilbert, 2009). In this study, participants are given various exercises to develop their soothing system, and help them to balance overactive threat.

SUMMARY:
The goal of this case series is to investigate whether a brief compassion-focused intervention is a safe, acceptable and feasible therapy for clients with bipolar affective disorder. The secondary questions are whether a brief compassion focused intervention for BPD clients is associated with changes in bipolar mood symptoms and/ or with changes in psychological processes linked to mood symptoms in bipolar, including: Self-compassion, perfectionism, social comparison and social safeness. Four visual analogue scales will also be completed daily by each participant throughout the project. These scales will measure domains relevant to BPAD symptomology and self-compassion.

Participants will complete a 4 session Compassion-Focused Therapy Intervention. The first session will involve completion of the psychoeducation and formulation work which was started during the initial assessment session. Each intervention session will also involve the introduction and practice of CFT techniques or exercises. The trial therapist will introduce the exercise and practice it together with the participant during the session. Participants will then be asked to continue practicing the exercises for homework. Their experience of the practice and any difficulties can then be discussed at the start of the next session.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older)
* Diagnosis of Bipolar Affective Disorder

Exclusion Criteria:

* Client considered to be actively at acute risk - judgement made by responsible clinical team and also by risk assessment at our first assessment session. High risk clients are excluded as due to time constraints it will be difficult to address risk issues and complete the intervention in the short time frame we have outlined.
* Client already receiving some form of CFT intervention, as this be a potential confounder.
* Level of English not strong enough to complete assessment and intervention sessions without use of interpreter. Again, due to time constraints it would be difficult to complete the intervention with clients in the timeframe outline whilst using an interpreter or navigating the language barrier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-06-09 (Estimated); Study Completion 2023-06-09 (Estimated)

PRIMARY OUTCOMES:
the Credibility and Expectancy Questionnaire (CEQ)(Devilly & Borkovec, 2000) | Assessment/Baseline Only
Client Satisfaction Questionnaire (CSQ-8) (Larsen, Attkison, Hargreaves & Nguyen, 1979). | Follow-up (2 weeks post-intervention)

SECONDARY OUTCOMES:
internal states scale (ISS) (Bauer, 1991) | Assessment (Baseline) and Follow-Up (2 weeks post intervention)
The Self Compassion Scale Short Form(SCS-SF) (Raes, Pommier, Neff & Van Gucht, 2011) | Assessment (Baseline) and Follow-Up (2 weeks post intervention)
The Short Revised Almost Perfect Scale (SAPS) (Rice, Richardson & Tueller, 2014) | Assessment (Baseline) and Follow-Up (2 weeks post intervention)
The Social Comparison Scale (Allan & Gilbert, 1995) | Assessment (Baseline) and Follow-Up (2 weeks post intervention)
The Social Safeness and Pleasure Scale (Gilbert et al, 2009) | Assessment (Baseline) and Follow-Up (2 weeks post intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry, Psychology & Neuroscience, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share individual data with researchers outside of research team at this time